CLINICAL TRIAL: NCT00695578
Title: A Randomized Right/Left Clinical Trial to Evaluate the Use of Biafine Cream Versus Standard Care in Subjects With Actinic Keratosis Post Cryotherapy
Brief Title: Clinical Trial to Evaluate Biafine Cream Versus Standard Care in Subjects With Actinic Keratosis Post Cryotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00000341; 31335 (Other: WakeForest)
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-07

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Biafine; bacitracin, polymyxin B drug combination; Bacitracin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biafin on left arm (Experimental): Subjects were randomized to apply Biafine® to wounds on the left forearm and polysporin (standard of care) to wounds on the right forearm. Medications were applied three times a day for 4 weeks to the areas that have been treated with liquid nitrogen at the baseline visit.
  Interventions: Drug: Biafine; Drug: Polysporin
- Biafin on right arm (Experimental): Subjects were randomized to apply Biafine to wounds on the right forearm and Polysporin to wounds on the left forearm. Medications were applied three times a day for 4 weeks to the areas that have been treated with liquid nitrogen at the baseline visit.
  Interventions: Drug: Biafine; Drug: Polysporin

INTERVENTIONS:
Drug: Biafine — Apply to wounds 3 times daily for 4 weeks: ingredients: purified water, liquid paraffin, glycol monostearate, stearic acid, propylene glycol, paraffin wax, squalene, avocado oil, trolamine sodium alginate, cetyl palmitate, methylparaben, sorbic acid, propyl paraben and fragrance.
Drug: Polysporin — over the counter Polysporin ointment 3 times daily for 4 weeks to wounds
  Other Names: Bacitracin

SUMMARY:
The purpose of this research study is to evaluate the use of Biafine Cream on wounds created by removal of actinic keratosis using cryotherapy in a clinical setting.

DETAILED DESCRIPTION:
Subjects were randomized to apply Biafine® to wounds on one forearm and polysporin (standard of care) to wounds on the other. Medications were applied three times a day for 4 weeks to the areas that have been treated with cryotherapy at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject must give written consent.
* Subjects must be >50 years of age, male or female.
* Subjects must have had cryotherapy treatment of at least one AK's on each forearm in the Dermatology Clinic.

Exclusion Criteria:

* Subjects age <50 years of age.
* Subjects with known allergy or sensitivity to topical Biafine or polysporin ointment.
* Inability to complete all study-related visits.
* Introduction of any other prescription medication, topical or systemic, for AK while participating in the study.
* Subjects using other topical agent's glycolic acid products, alpha-hydroxy acid products, retinoids and chemical peel agents in the treatment areas while on study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Biafin on Left: Subjects were randomized to apply Biafine® to wounds on the left forearm and polysporin (standard of care) to wounds on the right forearm. Medications were applied three times a day for 4 weeks to the areas that have been treated with liquid nitrogen at the baseline visit.
  Biafine: Apply to wounds 3 times daily for 4 weeks: ingredients: purified water, liquid paraffin, glycol monostearate, stearic acid, propylene glycol, paraffin wax, squalene, avocado oil, trolamine sodium alginate, cetyl palmitate, methylparaben, sorbic acid, propyl paraben and fragrance.
  Polysporin: over the counter Polysporin ointment 3 times daily for 4 weeks to wounds
- Biafin on Right: Subjects were randomized to apply Biafine® to wounds on the right forearm and polysporin (standard of care) to wounds on the left forearm. Medications were applied three times a day for 4 weeks to the areas that have been treated with liquid nitrogen at the baseline visit.
  Biafine: Apply to wounds 3 times daily for 4 weeks: ingredients: purified water, liquid paraffin, glycol monostearate, stearic acid, propylene glycol, paraffin wax, squalene, avocado oil, trolamine sodium alginate, cetyl palmitate, methylparaben, sorbic acid, propyl paraben and fragrance.
  Polysporin: over the counter Polysporin ointment 3 times daily for 4 weeks to wounds
Period: Overall Study
Arm/Group | Biafin on Left | Biafin on Right
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biafin on Left | Biafin on Right | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Severity Score
Description: The change in the Mean Severity Score from Baseline to Week 4 (or end of treatment) as measured by the Mean Combined Severity Scores for Erythema, Scab, and Thickness on a scale of 0-4 with 0=None 1=slight 2=mild 3= moderate 4= severe
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biafine Treatment Group: This group includes the forearm of the subjects that was randomized to apply Biafine® to wounds (either the left forearm or right forearm). Biafine was applied three times a day for 4 weeks to the areas that have been treated with liquid nitrogen at the baseline visit.
  Drug: Biafine Apply to wounds 3 times daily for 4 weeks: ingredients: purified water, liquid paraffin, glycol monostearate, stearic acid, propylene glycol, paraffin wax, squalene, avocado oil, trolamine sodium alginate, cetyl palmitate, methylparaben, sorbic acid, propyl paraben and fragrance.
  Other Names:
  • Biafine
- Polysporin Treatment Group: This group includes the forearm of the subjects that was randomized to apply Polysporin (standard of care) to wounds (either the left forearm or right forearm). Polysporin was applied three times a day for 4 weeks to the areas that have been treated with liquid nitrogen at the baseline visit.
  Drug: Polysporin over the counter Polysporin ointment 3 times daily for 4 weeks to wounds
  Other Names:
  • Bacitracin
Arm/Group | Biafine Treatment Group | Polysporin Treatment Group
Number analyzed (Participants) | 20 | 20
units on a scale | -1.52 (0.67) | -1.80 (1.44)

ADVERSE EVENTS:
Groups:
- Biafin Treatment Group: Experimental: Biafine Treatment Group
  This group includes the forearm of the subjects that was randomized to apply Biafine® to wounds (either the left forearm or right forearm). Biafine was applied three times a day for 4 weeks to the areas that have been treated with liquid nitrogen at the baseline visit.
  Drug: Biafine Apply to wounds 3 times daily for 4 weeks: ingredients: purified water, liquid paraffin, glycol monostearate, stearic acid, propylene glycol, paraffin wax, squalene, avocado oil, trolamine sodium alginate, cetyl palmitate, methylparaben, sorbic acid, propyl paraben and fragrance.
  Other Names:
  • Biafine
- Polysporin Treatment Group: Active Comparator: Polysporin Treatment Group
  This group includes the forearm of the subjects that was randomized to apply Polysporin (standard of care) to wounds (either the left forearm or right forearm). Polysporin was applied three times a day for 4 weeks to the areas that have been treated with liquid nitrogen at the baseline visit.
  Drug: Polysporin over the counter Polysporin ointment 3 times daily for 4 weeks to wounds
  Other Names:
  • Bacitracin
Arm/Group | Biafin Treatment Group | Polysporin Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes